CLINICAL TRIAL: NCT02201368
Title: Study to Evaluate the Effectiveness of Dietary Treatment With Triheptanoin in Patients With Long-chain Fatty Acid Beta-oxidation Defects
Brief Title: Triheptanoin Treatment Trial for Patients With Long-chain Fatty Acid Beta-oxidation Defects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: IMP management difficulties
Sponsor: Maria Luz Couce Pico (Other)
Collaborators: Fundación Ramón Domínguez (Other)
Responsible Party: Sponsor-Investigator, Maria Luz Couce Pico, MD, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2007/084; 2007-005578-29 (EudraCT Number)
Record Dates: First submitted 2013-03-22; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Long-chain Fatty Acid Transport Deficiency
Keywords: Triglycerides; Lipid Metabolism; Fatty Acids.
MeSH Terms: interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triheptanoin (Experimental)
  Interventions: Drug: Triheptanoin (SpezialölÒ 107®); Dietary Supplement: MCT (Medium-Chain Triglycerides)
- MCT (Medium-Chain Triglycerides) (Active Comparator)
  Interventions: Drug: Triheptanoin (SpezialölÒ 107®); Dietary Supplement: MCT (Medium-Chain Triglycerides)

INTERVENTIONS:
Drug: Triheptanoin (SpezialölÒ 107®) — * Randomization: Treatment with Triheptanoin for 6 months
  * Washout Period: Treatment with MCT(Medium-Chain Triglycerides)for 2 months
  * Crossover: Treatment with MCT(Medium-Chain Triglycerides)for 6 months
Dietary Supplement: MCT (Medium-Chain Triglycerides) — * Randomization: Treatment with MCT(Medium-Chain Triglycerides)for 6 months
  * Washout Period: Treatment with MCT(Medium-Chain Triglycerides)for 2 months
  * Crossover: Treatment with Triheptanoin for 6 months

SUMMARY:
The purpose of this study is to determine if administration Triheptanoin is an effective treatment for defects of the long-chain fatty acid beta-oxidation in young adults or adults. Period of treatment and follow-up will be 16 months.

DETAILED DESCRIPTION:
Triheptanoin treatment, in patients with long-chain fatty acid beta-oxidation defects, could cause not only a great improvement in their quality of life, also could prevent life-threatening signs, reducing symptoms and serious complications of their disease, like cardiomyopathy, Reye-like syndrome episodes and rhabdomyolysis. This result would occur by the effect of propionyl CoA primer on the Krebs cycle and, at the same time, would produce a gluconeogenic effect.

This treatment opens the door to be used in other diseases such as pyruvate carboxylase deficiency, glycogen storage disease and other diseases with energy problems.

All patients will be followed up until 16 months.

ELIGIBILITY:
Inclusion Criteria:

All patients with any of the following conditions:

* Long-chain 3-hydroxyacyl-coenzyme A dehydrogenase deficiency (LCHAD).
* Very long-chain acyl-coenzyme A dehydrogenase deficiency (VLCAD.)
* Mitochondrial trifunctional protein (MTP).
* Carnitine palmitoyltransferase I deficiency (CPT I).
* Carnitine Palmitoyltransferase II (CPT II).
* Carnitine-acylcarnitine translocase deficiency (CACT).

Positive skin biopsy: patients were deemed to commence the dietary treatment with Triheptanoin after evaluating the individual response in vitro in cultured fibroblasts. This response is based on the measurement of the production of propionyl-CoA, the incubation with fatty acids odd-chain, compared with control group fibroblasts.

The informed consent must be signed by the patient or family, in the case of minors.

Exclusion Criteria:

* No patient/family collaboration or the application of dietary treatment.
* No in vitro test response.
* Do not meet the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of metabolic decompensation. | up to 16 months
  This is a combined endpoint, including the number and/or severity of episodes of hypoglycemia, rhabdomyolysis, cardiomyopathy and liver failure after starting treatment with trihepatnoin.

SECONDARY OUTCOMES:
Differences in the profiles of acylcarnitines with control. | 6 months and 6 months in each arm treatment
Average values of transaminase and creatin kinase. | 6 months and 6 months in each arm treatment
Differences in the fatty acid composition of plasma and red blood cells. | 6 months and 6 months in each arm treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mª Luz Couce Pico, Study Chair — Hospital Clínico Universitario de Santiago; Jaume Campistol Plana, Principal Investigator — Hospital Sant Joan de Déu. Barcelona; Mercedes Martínez-Pardo, Principal Investigator — Hospital Universitario Ramon y Cajal; Mónica Ruiz Pons, Principal Investigator — Hospital Clínico Universitario Ntra. Sra. de Candelaria. Tenerife; Mª Teresa García Silva, Principal Investigator — Hospital 12 de Octubre. Madrid; Pablo Sanjurjo, Principal Investigator — Hospital de Cruces de Baracaldo - Bilbao; Koldo Aldamiz, Principal Investigator — Hospital de Cruces de Baracaldo - Bilbao; Inmaculada García Jiménez, Principal Investigator — Hospital Universitario Miguel Servet, Zaragoza
Locations (1):
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, Spain